CLINICAL TRIAL: NCT01906593
Title: A Post-marketing Study to Monitor the Safety of Beijing Tiantan Biological's Influenza Virus Vaccine Administered in Chinese Subjects Aged 60 Years or Older
Brief Title: A Post-marketing Safety Study of Beijing Tiantan Biological's Influenza Virus Vaccine in Elderly
Status: Completed | Type: Observational
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Beijing Tiantan Biological Products Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wu Jiang, Beijing Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, China
Other Study IDs: BJCDCWJ201301
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-03

CONDITIONS: Influenza; Vaccination Adverse Event
Keywords: safety; influenza vaccine; post-marketing
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Ecologic or Community
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tiantan biologial's vaccine: Tiantan Biological's vaccine group is the population injected with this vaccine.
- other group: Other vaccine group is the population injected with other manufacturers' vaccine except Tiantan Biological CO, Ltd.

SUMMARY:
To monitor the safety of Beijing Tiantan Biological's influenza vaccine in elderly through Adverse Events Following Immunization Surveillance System of China.

The hypothesis is that there is no significant difference in the occurrence of adverse events among influenza vaccines manufactured by independent companies.

DETAILED DESCRIPTION:
In 2011 and 2012, Beijing Municipal Health Bureau launched the free influenza vaccination campaign among children aged 6-18 years old and the elderly aged 60 years old and above. Inactivated split-virion vaccines from Beijing Tiantan Biological Products Company were used for the elderly in the campaign.

All vaccine recipients provided written informed consent, containing information about the vaccine, possible adverse effects, and medical care.

Adverse events were collected through the National Immunization Information System's National Adverse Events Following Immunization (AEFI) Surveillance System, which was established in 2005 on the basis of World Health Organization (WHO) guidelines. According to the Guideline for the Identification of Adverse Reaction after Immunization issued by the Chinese Ministry of Health in 2008, Beijing CDC and local prefectural CDC must organize an expert panel to investigate adverse events and assess causality, using criteria based on Chinese Standard Procedures for Vaccination. The panels consist of physicians, epidemiologists, pharmacists, and other relevant experts. In general, expert panels investigate deaths, life-threatening illnesses, and permanent disabilities, and immunization-program managers or vaccination providers investigate common, minor adverse events. Adverse events are classified into one of five categories: vaccine reactions (common and minor to rare and more serious), program errors, coincidental illnesses, psychogenic reactions, and unclassifiable events.

At the time of vaccination, vaccinees were instructed to report any adverse event to physicians or vaccination providers. Adverse events that were fatal or that resulted in disability and clusters of events (i.e., notably high numbers of similar adverse events related to a certain vaccine) were required to be reported within 2 hours after their occurrence. The following adverse events were required to be reported within 2 days after their occurrence: anaphylaxis or other allergic reactions occurring within 24 hours after vaccination; fever (axillary temperature, >37.5°C), angioedema, or a local injection-site reaction (diameter, >2.5 cm) occurring within 5 days after vaccination; purpura, an Arthus reaction, febrile convulsion, seizure, or polyneuritis occurring within 15 days after vaccination; and the Guillain-Barré syndrome occurring within 3 months after vaccination. Other reactions that were common and minor (e.g., mild pain and fatigue) were not required to be reported.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 60 years and above on the day of immunization, who are eligible for seasonal influenza vaccination.
2. In the judgement of the study doctor are determined to be in reasonable health considering their age and able to comply with all study procedure.

Exclusion Criteria:

1. History of any serious reaction to flu vaccine, or any materials in the vaccine, and to eggs (including ovalbumin) and chicken protein.
2. Receipt of a live vaccine within 4 weeks prior to Study Day 1.
3. Any condition, which in the opinion of the study doctor, might interfere with the evaluation of the study objective.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Beijing subjects aged 60 years or older, at the time of routine visit to a participating clinic or hospital for annual influenza vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 536812 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
the rate of reported adverse events | 3 months after vaccination
  The rate of reported adverse events was calculated by dividing the number of vaccinees who reported having an event by the number of vaccine doses administered. The cumulative rate of reported adverse events was calculated by dividing the number of vaccinees who reported having an event by the number of vaccine doses administered from the beginning of the first week to the end of each week.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, Master, Principal Investigator — Beijing Centers for Disease Prevention and Control, China